CLINICAL TRIAL: NCT00474214
Title: Safety And Feasibility of Early DischargE - a Prospective And Randomized Trial of Low-risk Primary PCI Patients (The SAFE-DEPART Trial)
Brief Title: Safety And Feasibility of Early DischargE - a Prospective And Randomized Trial of Low-risk Primary Percutaneous Coronary Intervention (PCI) Patients
Acronym: SAFE-DEPART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: McMaster University (Other); Regional Medical Associates Research Scholarship Fund (Unknown)
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 06-387
Record Dates: First submitted 2007-05-15; First posted 2007-05-16 (Estimated); Last update posted 2010-02-23 (Estimated); Status verified 2010-02

CONDITIONS: Myocardial Infarction
Keywords: STEMI; Primary PCI; Length of Stay; Early Discharge
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Early hospital discharge facilitated by close nurse practitioner follow-up

SUMMARY:
The purpose of this study is to determine if early hospital discharge (at 48-72 hours), is feasible, safe, cost-effective, and/or improves compliance with medications, positive lifestyle changes and quality-of-life, in low-risk patients with ST-elevation myocardial infarction treated with primary percutaneous coronary intervention (primary PCI).

DETAILED DESCRIPTION:
Patients with acute ST-segment elevation myocardial infarction (STEMI) have traditionally been hospitalized for at least 5-7 days to monitor for serious complications, including heart failure, arrhythmias, re-infarction and death. With the advent of primary percutaneous coronary intervention (PCI) as the treatment of choice for STEMI, fewer patients are completing their infarcts and the incidence of complications is decreasing. The Zwolle Primary PCI Index is one of several externally validated risk scores that can be used to identify low-risk primary PCI patients who can safely be discharged at 48-72 hours. Recent reviews have found that a majority of primary PCI patients with risk scores that deem them "low-risk" are kept in hospital longer than predicted by these scores.

SAFE-DEPART is a trial where low-risk primary and rescue PCI patients will be randomized either to an intervention arm (early hospital discharge, early outpatient follow-up with a nurse practitioner) or to standard of care (no recommended discharge date, no outpatient follow-up with a nurse practitioner). At 6 weeks time, a blinded research assistant will contact patients and collect data on feasibility, safety, quality-of-life, and cost-effectiveness outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patient with ST-elevation myocardial infarction (STEMI)
* Treatment with either primary or rescue PCI
* Zwolle risk score <= 3

Exclusion Criteria:

* Developed MI while in hospital for another reason
* Time from angioplasty to enrollment > 24 hours

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2007-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Safety: All-cause mortality | 6 weeks
Safety: Readmission for any of CHF, unstable angina, arrhythmia, re-infarction, revascularization, stroke, or major bleeding requiring transfusion | 6 weeks
Feasibility: Proportion of patients in the intervention group discharged within 72 hours ("feasible" if >= 70%)
Feasibility: Proportion of patients in the intervention group who saw nurse practitioner within 3 days of discharge ("feasible" if >= 80%)
Feasibility: Proportion of patients in the intervention group who saw nurse practitioner within 5 days of discharge ("feasible" if >= 90%)

SECONDARY OUTCOMES:
Quality of life, as measured by the SF-36 questionnaire | 6 weeks
Compliance with medications | 6 weeks
Compliance with smoking cessation | 6 weeks
Attendance at first cardiac rehabilitation session | 6 weeks
Cost-effectiveness | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Kotowycz, MD, MBA, Principal Investigator — McMaster University; Madhu K Natarajan, MD, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- Hamilton Health Sciences, Hamilton, Ontario, Canada

REFERENCES:
- [Result] Kotowycz MA, Cosman TL, Tartaglia C, Afzal R, Syal RP, Natarajan MK. Safety and feasibility of early hospital discharge in ST-segment elevation myocardial infarction--a prospective and randomized trial in low-risk primary percutaneous coronary intervention patients (the Safe-Depart Trial). Am Heart J. 2010 Jan;159(1):117.e1-6. doi: 10.1016/j.ahj.2009.10.024. PMID 20102876